CLINICAL TRIAL: NCT05073926
Title: Acquisition and Persistence of Rifampicin Resistance in Staphylococcus Aureus During and After Treatment for Latent Tuberculosis
Brief Title: Rifampicin Resistance in S. Aureus During and After Treatment for Latent Tuberculosis
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Anton Reepalu, Principal Investigator, Region Skane
Other Study IDs: 2021-02312
Record Dates: First submitted 2021-09-09; First posted 2021-10-12 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Latent Tuberculosis; Staphylococcus Aureus
Keywords: rifampicin; isoniazide; staphylococcus aureus; latent tuberculosis; Drug Resistance, Microbial
MeSH Terms: conditions — Latent Tuberculosis; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Persons with latent tuberculosis treated with 4 months rifampicin: Oral rifampicin 10 mg/kg (max 600mg) once daily during 4 months
  Interventions: Other: No intervention is part of the study protocol
- Persons with latent tuberculosis treated with 6-9 months isoniazide: Oral isoniazide 5 mg/kg (max 300mg) once daily in combination with 40mg vitamin B6 (pyridoxin) during 6-9 months
  Interventions: Other: No intervention is part of the study protocol

INTERVENTIONS:
Other: No intervention is part of the study protocol — No intervention is part of the study protocol. The choice of treatment for latent tuberculosis is is made by the treating physician.

SUMMARY:
Two commonly used treatments for latent tuberculosis infection are either 4 months rifampicin or 6-9 months isoniazid. The invistigators will study the risk of acquisition of rifampicin resistance in commensal Staphylococcus aureus in persons treated with rifampicin versus in persons treated with isoniazide. Through repeated swab cultures before, during, and after treatment the investigators will also investigate potential accumulation of mutations associated with rifampicin resistance over time. Finally, household contacts to persons with rifampicin-resistant S. aureus will be examined to investigate whether onward transmission of rifampicin-resistant S. aureus occurs within households.

DETAILED DESCRIPTION:
The use of rifampicin for treatment of latent tuberculosis has gained popularity due to a shorter treatment course compared with isoniazide (4 versus 6-9 months) since this can lead to a higher proportion of treatment completion. An estimated 25% of the global population is latently infected with tuberculosis. Hence, a shift towards rifampicin instead of isoniazide, which has a more narrow antibacterial spectrum, could have a large impact on the prevalence of rifampicin resistance among commensal bacteria with pathogenic potential, such as Staphylococcus aureus (S.aureus).

The investigators will investigate the risk of acquisition of rifampicin resistance in commensal S.aureus during out-patient treatment for latent tuberculosis using 4 months rifampicin versus 6-9 months isoniazide at Skåne University Hospital in Malmö, Sweden.

Swabs will be obtained from the nose, throat, groin and possible wounds for culture and resistance testing before, during and after cessation of treatment for latent tuberculosis. Whole genome sequencing will be used to analyze accumulation of mutations over time and to determine if it is the primarily detected S.aureus that develop resistance or if the individual is colonized by new, rifampicin-resistant S.aureus over the course of treatment. Household contacts to persons with rifampicin-resistant S.aureus will be examined to investigate onward spread of bacteria within a household.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with latent tuberculosis
* prescribed either 4 months rifampicin or 6-9 months isoniazide
* informed consent

Exclusion Criteria:

* none

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals 16 years or older diagnosed with latent tuberculosis and prescribed prophylactic treatment with rifampicin or isoniazide as part of routine care at the out-patient department of the departments for infectious diseases at Skåne University Hospital in Malmö, Helsingborg and Växjö, Sweden.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of rifampicin resistant S. aureus in individuals treated with rifampicin versus isoniazide for latent tuberculosis infection | 5 months
  The proportion of individuals colonized with rifampicin-resistant S.aureus during and after 4 months treatment with rifampicin for latent tuberculosis will be compared with a control group of individuals treated with isoniazide during a similar time period to determine the relative risk of acquiring rifampicin-resistant S.aureus carriage.

SECONDARY OUTCOMES:
Frequency of mutations associated with rifampicin resistance in S.aureus during and after rifampicin treatment for latent tuberculosis infection | 10 months
  The frequency of mutations associated with rifampicin resistance will be determined thorugh whole-genome sequencing at pre-specified time points before, during and after 4 months treatment with rifampicin for latent tubeculosis infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No